CLINICAL TRIAL: NCT05380349
Title: A Phase 1 Study of Combination Drug Therapy Based on Personalized Cancer Stem Cell (CSC) High-Throughput Drug Screening (HTS) With Standard of Care for Newly Diagnosed Glioblastoma
Brief Title: Personalized Cancer Stem Cell High-Throughput Drug Screening for Glioblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 161581
Record Dates: First submitted 2022-04-21; First posted 2022-05-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Newly Diagnosed Glioblastoma

STUDY DESIGN:
Intervention Model Description: single-center Phase 1 open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized Combination Drug Therapy for Cancer Stem Cells (Experimental): Administer combinations of up to 3 FDA approved drugs from a panel of compounds selected based on high throughput screening
  Interventions: Drug: combinations of up to 3 FDA approved drugs from a panel of compounds

INTERVENTIONS:
Drug: combinations of up to 3 FDA approved drugs from a panel of compounds — personalized drug combinations

SUMMARY:
Proposed treatment of subjects with newly diagnosed glioblastoma with novel personalized drug regimens identified to be effective in vitro using cancer stem cells derived from their individual tumors, alongside standard of care radiation and TMZ.

DETAILED DESCRIPTION:
A panel of FDA approved drugs will be tested by high throughput screening, which is CLIA certified allowing for clinical decisions based on the results, to identify a combination of up to 3 drug candidates for treating individual patients. Lead candidates will be evaluated by pharmacists and a team of physicians, to confirm that prescribed drugs do not utilize pharmacological/ metabolic pathways that are known to increase the likelihood of toxicity, prior to initiating treatment. Investigational drug therapy, targeting CSCs, will be initiated alongside standard of care chemoradiation with TMZ.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of GBM (WHO grade 4)
* Subjects ≥18 years of age
* Patients must have a life expectancy of >6 months
* Patients must have a surgically accessible tumor with the intent for a gross or near total resection of the tumor mass (GBM, WHO grade 4)
* Patients must have a KPS rating of ≥70
* Patients should not have received any prior systemic anti-cancer therapy
* Patients must be negative for HIV, Hepatitis B and C
* Baseline hematologic studies and chemistry and coagulation profiles must meet the following criteria:

  * Hemoglobin (Hgb)> 8 g/dL
  * Absolute Neutrophil Count (ANC) > 1,000/mm3
  * Platelet count > 100,000/mm3
  * Creatinine < 2 mg/dL
  * Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) < 3x upper limit of normal (ULN)

Exclusion Criteria:

* Metastatic disease
* Diseases or conditions that obscure toxicity or dangerously alter drug metabolism
* Serious intercurrent medical illness
* Inadequately controlled hypertension
* History of myocardial infarction or unstable angina within 6 months
* History of stroke or transient ischemic attack within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
determine safety of CSC/HTS-based combination drug therapy | From date of first dose of investigational drug regimen until date of first documented progression or death from any cause, whichever came first, assessed up to 24 months.
  incidence of treatment-related AEs, laboratory abnormalities, and SAEs as assessed by CTCAE version 5.0

SECONDARY OUTCOMES:
Efficacy of CSC/HTS-based combination drug therapy | From inclusion in the study up to approximately 36 months
  Response assessment per Response Assessment in Neuro-Oncology (RANO) criteria
Efficacy of CSC/HTS-based combination drug therapy | From inclusion in the study until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 36 months
  Progression-free survival (PFS)
Efficacy of CSC/HTS-based combination drug therapy | From inclusion in the study until date of death from any cause, assessed up to approximately 36 months
  Median overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cobbs, Principal Investigator — Ivy Center for Advanced Brain Tumor Treatment
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No